CLINICAL TRIAL: NCT02680457
Title: Effect of the Administration of Insulin Degludec Versus Insulin Glargine on Glycemic Variability in Patients With Type 2 Diabetes Mellitus Drug-naïve
Brief Title: Effect of Insulin Degludec Versus Insulin Glargine on Glycemic Variability in Patients With Type 2 Diabetes Mellitus
Acronym: Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, PhD, University of Guadalajara
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CT-DG-140282-JLRN
Record Dates: First submitted 2015-12-07; First posted 2016-02-11 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Degludec - Insulin Glargine (Active Comparator): Insulin Degludec 10 IU SC every 24 hours for 6 days Washout for 14 days Insulin Glargine 10 IU SC every 24 hours for 6 days
  Interventions: Drug: Insulin Degludec; Drug: Insulin Glargine
- Insulin Glargine - Insulin Degludec (Active Comparator): Insulin Glargine 10 IU SC every 24 hours for 6 days Washout for 14 days Insulin Degludec 10 IU SC every 24 hours for 6 days
  Interventions: Drug: Insulin Degludec; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Degludec — Insulin Degludec 10 IU SC every 24 hours for 6 days
  Other Names: Tresiba ® (Novo Nordisk A/S. Bagsvaerd, Denmark)
Drug: Insulin Glargine — Insulin Glargine 10 IU SC every 24 hours for 6 days
  Other Names: Lantus ® (Sanofi-Aventis Deutschland GmbH. Frankfurt, Germany)

SUMMARY:
Type 2 diabetes mellitus (T2DM) is characterized by wide fluctuations of glucose. The long-acting insulin has showed to improve glycemic variability however the behavior of insulin glargine versus insulin degludec is unknown.

DETAILED DESCRIPTION:
Cross-over, double dummy, randomized, clinical trial was carried out. The sample size was calculated using the formula for clinical trials of mean differences with an "n" of 6 patients per group was obtained. Patients between 30 and 65 years of age will be included with T2DM, without hyperglycemic drugs, hemoglobin A1c (A1C) 6.5 to 11.0 % and with written signature consent. They were assigned randomly by sealed envelope either to received insulin Degludec (Novo Nordisk A/S. Bagsvaerd, Denmark) or insulin Glargine (Sanofi-Aventis Deutschland GmbH. Frankfurt, Germany) [10 international units (IU) subcutaneous (SC) every 24 hours for six days], patients who were administered initially insulin Degludec corresponded then insulin Glargine and vice versa, with a washout period of 14 days between each intervention.

The clinical findings and laboratory tests included a metabolic profile and biosafety, which will be made at baseline. Body weight, body mass index and blood pressure were performed during the initial visit, likewise, interstitial glucose concentrations by ambulatory continuous glucose monitoring system (Guardian®, Medtronic MiniMed, Northridge), through which the mean amplitude of glucose excursions (MAGE) and area under the curve of glucose were calculated, which served to assess the glycemic variability. Adverse events and adherence to treatment are documented. Statistical analysis: Mann-Whitney U test, Chi2, Fisher exact test. It is considered with significance at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM without treatment for at least 3 months Body mass index (BMI) from 25.0-34.9 kg/m2 Diagnosis of T2DM
* Fasting plasma glucose ≤300 mg/dL at the time of scrutiny
* A1C between 6.5 and 11%
* Written informed consent

Exclusion Criteria:

* Women pregnant or breastfeeding
* Untreated thyroid disease and/or uncontrolled hypertension [≥150 systolic and diastolic ≥90]
* Consumption of oral agents or other medications or supplements with proven properties that modify the behavior of glucose. In the case of antihypertensives, these may be included if treatment was not modified previous 3 months and no change during the study.
* Total cholesterol >240 mg/dL
* Triglycerides ≥400 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) more than twice the normal range
* Glomerular filtration rate <60 mL/min [Cockcroft-Gault]

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of patients: 12 in a crossover intervention. Interventions: 2. Washout period before the cross-over intervention. Protocol violations were detected at the end of the study in patients of both groups
Groups:
- Insulin Degludec - Insulin Glargine: Insulin Degludec: 10 IU subcutaneous (SC) every 24 hours for 6 days Washout period for 14 days Insulin Glargine 10 IU SC every 24 hours for 6 days
- Insulin Glargine - Insulin Degludec: Insulin Glargine: 10 IU subcutaneous (SC) every 24 hours for 6 days Washout period for 14 days Insulin Degludec 10 IU SC every 24 hours for 6 days
Period: Initial Intervention
Arm/Group | Insulin Degludec - Insulin Glargine | Insulin Glargine - Insulin Degludec
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Insulin Degludec - Insulin Glargine | Insulin Glargine - Insulin Degludec
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Cross-over Intervention
Arm/Group | Insulin Degludec - Insulin Glargine | Insulin Glargine - Insulin Degludec
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Characteristics of the entire group
Groups:
- Insulin Total Group: Total Group of Patients with Type 2 Diabetes mellitus
Arm/Group | Insulin Total Group
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 80.5 (13.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (2.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 114.8 (8.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 75.8 (6.4)
Hemoglobin A1c [Mean (Standard Deviation); unit: % of Hemoglobin A1c] | 8.2 (1.4)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dl] | 181 (59.8)
Uric Acid [Mean (Standard Deviation); unit: mg/dl] | 4.6 (1.4)
Creatinine [Mean (Standard Deviation); unit: mg/dl] | 0.7 (0.2)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 174.8 (29.5)
High-density lipoprotein-cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dl] | 42.3 (9.4)
Low-density lipoprotein-cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dl] | 92.6 (27.9)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 199.3 (84.5)
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: mg/dl] | 25.8 (11.3)
Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: mg/dl] | 41.6 (25.9)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Variability: Mean Amplitude of Glucose Excursion (MAGE)
Description: Mean amplitude of interstitial glucose excursions (MAGE) during the last 48 h of the ambulatory continuous glucose monitoring of 3 days (Guardian®, Medtronic MiniMed, Northridge); starting in the day 3 of the administration of insulin degludec or glargine
Time Frame: 2 days
Population: Comparison between both interventions. There are not baseline values of this measurements due to a design error. There were technical problems with the measurements.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Insulin Degludec: Patients who received:
  Insulin Degludec: 10 IU SC every 24 hours for 6 days, from both arms of the study
- Insulin Glargine: Patients who received:
  Insulin Glargine: 10 IU SC every 24 hours for 6 days, from both arms of the study
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 12 | 12
mg/dl | 75.2 (38.9) | 68.5 (47.4)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine; Test type: Superiority; p = 0.630, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Glycemic Variability: Area Under the Curve of Glucose
Description: Area under the curve of glucose of the second day of continuous ambulatory glucose monitoring of 3 days (Guardian®, Medtronic MiniMed, Northridge)
Time Frame: Every 5 min for 24 hours on day 5 post-dose
Population: Area Under the Curve of Glucose in a patient (Insulin Degludec group) could not be calculated. There are not baseline values of this measurements due to a design error. There were technical problems with the measurements.
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 11 | 12
mg*h/dL | 46776 (17860) | 46499 (16971)
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the beginning of the study until a month after the end of the intervention for each patient, an average of 2 months
Groups:
- Insulin Degludec: Patients with Type 2 Diabetes mellitus
  Insulin Degludec: 10 IU SC every 24 hours for 6 days
- Insulin Glargine: Patients with Type 2 Diabetes mellitus
  Insulin Glargine: 10 IU SC every 24 hours for 6 days
Arm/Group | Insulin Degludec | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (N=12) | Insulin Glargine (N=12)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Lower limb paresthesias (Nervous system disorders) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mild hypoglycemia (Endocrine disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
There were technical problems with the measurement of the outcomes. Design errors and protocol violations were detected at the end of the study. Therefore, the results are considered unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes